CLINICAL TRIAL: NCT00943371
Title: A Double-Blind, Randomized, Placebo-Controlled, Single and Divided Rising-Dose, Sequential Panel Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of MK6349 in Subjects With Type 2 Diabetes
Brief Title: A Single-Dose Study of MK6349 in Patients With Type 2 Diabetes (6349-002)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 6349-002; MK6349-002; 2007_597
Record Dates: First submitted 2009-07-21; First posted 2009-07-22 (Estimated); Last update posted 2015-08-27 (Estimated); Status verified 2015-08

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental): MK6349
  Interventions: Drug: MK6349
- 2 (Placebo Comparator): Placebo to MK6349
  Interventions: Drug: Comparator: Placebo to MK6349

INTERVENTIONS:
Drug: MK6349 — Panel A: MK6349 in single doses beginning at 16 mg and rising to 90 mg in up to four treatment periods Panel B: MK6349 in single doses beginning at 90 mg and rising to 160 mg in up to four treatment periods Panel C: MK6349 in divided doses beginning at 20 mg q.a.c. (before each meal) and rising to 50 mg q.a.c. in up to four treatment periods
  Arms: 1
Drug: Comparator: Placebo to MK6349 — Panel A: Placebo to MK6349 in single doses in up to four treatment periods Panel B: Placebo to MK6349 in single doses in up to four treatment periods Panel C: MK6349 in divided doses q.a.c. (before each meal) in up to four treatment periods
  Arms: 2

SUMMARY:
A single dose study to assess the safety, tolerability, pharmacokinetics and pharmacokinetics of MK6349 in Type 2 Diabetics.

ELIGIBILITY:
Inclusion Criteria:

* Subject is a non-smoking male or female (females must be postmenopausal, had a tubal ligation or a hysterectomy) between 18 to 55 years of age
* Subject has Type 2 Diabetes and is currently being treated with diet and exercise alone or with less than 3 oral diabetes drugs

Exclusion Criteria:

* Subject is on insulin or a PPAR agonist medication
* Subject has Type 1 diabetes

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2007-08; Primary Completion 2007-09 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of MK6349 after single and divided rising doses based on assessment of clinical and laboratory evaluations and adverse experiences | Through 30 days after the last dose of study drug
15-Hour weighted mean plasma glucose (WMG) concentration | 15 hours postdose

SECONDARY OUTCOMES:
4-Hour weighted mean plasma glucose (WMG) concentration | 4 hours postdose

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC